CLINICAL TRIAL: NCT07347860
Title: Clinical Study of Recombinant Anti-CD19m-CD3 Antibody Injection (A-319) in the Treatment of Active Rheumatoid Arthritis
Brief Title: Clinical Study of (A-319) in the Treatment of Active Rheumatoid Arthritis
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: ITabMed Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Qiubai Li, Director, Head of Department of Rheumatology and Immunology, Principal Investigator, Professor, Wuhan Union Hospital, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHCT250824
Record Dates: First submitted 2025-08-19; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: Rheumatoid arthritis (RA); A-319
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A-319 subcutaneous intervention (Experimental): A-319 will be administered subcutaneously in two ascending dose levels: Dose A and Dose B, with a total treatment course of 4 weeks. Expected enrollment: Dose A, B: 3+N; Total: 12-18 participants
  Interventions: Biological: A-319

INTERVENTIONS:
Biological: A-319 — A-319 will be dosed according to the assigned group.

SUMMARY:
The primary objective of the study was to evaluate the safety and tolerability of A-319 in patients with active rheumatoid arthritis.

DETAILED DESCRIPTION:
Active rheumatoid arthritis (RA) is an autoimmune disease characterized by erosive arthritis as its primary clinical manifestation. A-319 is a recombinant CD19xCD3 bispecific antibody that activates T cells in vivo and targets and kills pathogenic B cells. A-319 is currently in clinical trials for B-cell hematologic malignancies. Preclinical results in animal models of systemic lupus erythematosus (SLE) and RA have also demonstrated that A-319 can alleviate or eliminate autoimmune disease-related symptoms and progression by depleting pathogenic B cells in individuals with autoimmune diseases. This investigator-initiated trial (IIT) evaluated the safety, tolerability, pharmacokinetic profile, biological markers, and preliminary efficacy of A-319 in the treatment of patients with rheumatoid arthritis (RA) who have refractory responses to at least two different therapies with different mechanisms of action.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years (inclusive), gender unrestricted.
2. Meet the 2010 American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) classification criteria, with a diagnosis of rheumatoid arthritis for at least 24 weeks.
3. Patients with rheumatoid arthritis who have previously responded inadequately to at least one csDMARD and who have not responded to 12 weeks of combined treatment with at least one bDMARD or/and tsDMARD with a different mechanism of action in addition to their original csDMARD, such as those with insignificant improvement in swollen/tender joints, physical condition, or disease activity.
4. Experiencing at least one of the following clinical manifestations suggestive of moderate to severe RA disease activity:

1) C-reactive protein-based 28-joint disease activity index (DAS28-CRP) >3.2 or clinical disease activity index (CDAI) >10; 2) Clinical manifestations and/or symptoms suggestive of disease activity, including acute inflammatory markers (ESR, CRP) and imaging findings, and joint-related or other symptoms. 5. At the screening and baseline visits, patients must have ≥ 6 tender joints (TJCs) per 68 units and ≥ 4 swollen joints (SJCs) per 66 units.

6. If the patient is taking oral glucocorticoids, the dose of prednisone or its equivalent must be ≤ 7.5 mg/day and maintained stable for at least 2 weeks before the first dose.

7. Patients must have voluntarily signed the informed consent form, communicated well with the investigator, and completed all visits as required by the protocol.

Exclusion Criteria:

Subjects with other autoimmune diseases that the investigator considers would not potentially benefit from A-319 treatment; or conditions that interfere with the assessment of joint swelling and pain. 2. Use of abatacept, infliximab, adalimumab, or tocilizumab within 6 weeks prior to the first treatment with the study drug; use of etanercept, anakinra, immune globulin, or blood products within 4 weeks prior to the first treatment with the study drug; or use of a JAK inhibitor (e.g., tofacitinib, baricitinib, or upadacitinib), mycophenolate mofetil, cyclosporine, or iguratimod within 2 weeks prior to the first treatment with the study drug.

3. Use of B-cell depleting therapy, such as rituximab, within 3 months prior to the first treatment with the study drug; cell counts must have returned to acceptable levels or baseline.

4. Subjects with any periprosthetic joint infection. 5. Patients with immunodeficiency (defined as immunoglobulin G ≤ 5g/L). 6. History of demyelinating diseases, including, but not limited to, multiple sclerosis, Guillain-Barré syndrome, and neuromyelitis optica (Devic's disease). 7. Laboratory values: Hemoglobin level < 9.0 g/dL, absolute white blood cell (WBC) count < 3.0 × 109/L (< 3000/mm3), or absolute neutrophil count < 1.2 × 109/L (< 1200/mm3), or absolute lymphocyte count < 0.8 × 109/L (< 800/mm3); thrombocytopenia, defined as a platelet count < 100 × 109/L (< 100,000/mm3); age-appropriate estimated glomerular filtration rate (eGFR) < 45 mL/min/1.73 m2, proteinuria ≥ 3+; total bilirubin (T-bili), aspartate aminotransferase (AST), and alanine aminotransferase (ALT) exceeding 1.5 times the upper limit of normal (ULN). 8. Receipt of live or live attenuated vaccines within 30 days prior to first medication use.

9. Active hepatitis during the screening period, or positive hepatitis B virus surface antigen (HBsAg), or positive hepatitis B virus core antibody (HBcAb) plus hepatitis B virus (HBV) deoxyribonucleic acid (DNA), or positive hepatitis C virus (HCV) antibody plus HCV RNA; history of human immunodeficiency virus (HIV) infection, or positive HIV antibody during the screening period; or positive Treponema pallidum antibody during the screening period.

10. Chronic active infection or acute infection requiring systemic treatment with antibiotics, antivirals, antiparasitics, or antifungals within 2 weeks prior to screening, or superficial skin infection requiring treatment within 1 week prior to screening (Note: Patients can be rescreened after the infection is resolved). 11. Major surgical procedure (craniotomy, thoracotomy, or laparotomy) or unhealed wounds, ulcers, or fractures within 4 weeks prior to the first dose of study drug, or plans for major surgery during the study.

12. A history of a major clinical illness (such as circulatory system disorders, endocrine system disorders, nervous system diseases, respiratory system diseases, hematologic diseases, immune system diseases, psychiatric disorders, and metabolic instability) that the investigator believes will pose a risk to the patient's safety, or that may affect safety or efficacy analysis if the disease/symptom worsens during the study. For example: Cardiovascular disease: history of acute myocardial infarction, unstable angina, or severe arrhythmias (multi-source frequent premature ventricular contractions, ventricular tachycardia, or ventricular fibrillation) within 6 months prior to screening; New York Heart Association (NYHA) class III-IV.

13. Possible active Mycobacterium tuberculosis infection, defined as: positive sputum smear/sputum culture within 3 months prior to screening/during the screening period, or chest X-ray (anteroposterior and lateral)/lung CT indicating active tuberculosis infection (tuberculosis testing will be performed according to the site's protocol if ethically required).

14. Subjects with a malignancy within 5 years prior to screening (excluding completely cured in situ cervical cancer, non-metastatic squamous cell carcinoma or basal cell carcinoma of the skin, ductal carcinoma in situ of the breast, and papillary thyroid carcinoma).

15. History of major organ transplant (e.g., heart, lung, kidney, liver) or hematopoietic stem cell/or bone marrow transplant).

16. Participation in any clinical trial within 4 weeks prior to the first dose of study drug or within 5 half-lives of the study drug in the clinical trial (whichever is longer, unless otherwise specified).

17. Patients undergoing acute or consolidation medication for depression and experiencing suicidal thoughts within 6 months. 18. Women who are pregnant or breastfeeding, or who plan to become pregnant or breastfeed during the study; or men whose partners plan to become pregnant during the study.

19. Any reason that the researcher deems would prevent the subject from participating in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-01-08 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | Time frame: Within 1 year after subcutaneous injection of A-319
  Safety and tolerability will be assessed by incidence and severity of adverse events (AEs) and serious AEs (SAEs)

SECONDARY OUTCOMES:
Pharmacokinetics of A-319 | Within 1 month after subcutaneous injection of A-319
  Blood samples were collected from the sampling points according to the plan, and the concentration of A-319 in the patients' serum was measured and the pharmacokinetic parameters were calculated
Numbers of Participants with positive antidrug antibodies in peripheral blood | Before dosing on day 1, before dosing on day 15, on days 28-29, and at weeks 8, 16, and 24
  To evaluate immunogenicity of A-319
Pharmacodynamics of A-319 | Within 1 month after subcutaneous injection of A-319
  Pharmacodynamics will be assessed by levels of cytokines (IL-6, IL-8, IL-10, IFN-γ, TNF-α) in peripheral blood
Pharmacodynamics of A-319 | Within 1 month after subcutaneous injection of A-319
  Pharmacodynamics will be assessed by levels of lymphocyte subsets in peripheral blood

OTHER OUTCOMES:
68 swollen joints and 66 tender joints assessed | A-319 within 1 year after subcutaneous injection (Day 15, Day 28, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12)
  68 swollen joints and 66 tender joints were assessed by independent joint assessors and reviewed by safety assessors.
Physician's Global Assessment of Disease (PhGADA-VAS) | A-319 within 1 year after subcutaneous injection (Day 15, Day 28, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12)
  The PhGADA_VAS is a component of the ACR evaluation and is used to assess treatment efficacy.
  The PhGADA_VAS uses a visual analog scale (0-100 mm, with 0 indicating no disease activity and 100 indicating very severe disease activity) to assess a patient's current disease activity.
Disease activity score based on C-reactive protein (DAS28-CRP) | A-319 within 1 year after subcutaneous injection (Day 15, Day 28, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12)
  The DAS28-CRP score includes the following: swollen joints, tender joints, CRP, PhGADA_VAS
Disease activity score based on erythrocyte sedimentation rate (DAS28-ESR) | A-319 within 1 year after subcutaneous injection (Day 15, Day 28, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12)
  The DAS28-ESR score includes the following: swollen joints, tender joints, ESR, PhGADA_VAS swelling degree, and pain degree.
American College of Rheumatology criteria 20, 50, and 70 (ACR20, ACR50, ACR70) | A-319 within 1 year after subcutaneous injection (Day 15, Day 28, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12)
  ACR20 is defined as an improvement of at least 20% in the ACR score. ACR50 and ACR70 are defined as improvements of at least 50% and 70% in the ACR score. That is, an improvement of at least 20%, 50%, and 70%
Patient Global Assessment of Disease (PhGA-VAS) | A-319 within 1 year after subcutaneous injection (Day 15, Day 28, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12)
  PhGA_VAS is a component of the ACR evaluation and is used to assess efficacy.The PhGA_VAS assesses the patient's overall assessment of their current illness using a visual analog scale (0-100 mm, with 0 indicating very good and 100 indicating very poor). It asks the patient how they feel about their current illness.
Patient's global assessment of joint pain (VAS) | A-319 within 1 year after subcutaneous injection (Day 15, Day 28, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12)
  The patient's global assessment of joint pain (VAS) is a component of the ACR evaluation and is also used to assess efficacy. PhGADA_VA has only a single question, which asks patients, "How severe is the joint pain caused by rheumatoid arthritis?" The assessment is done using a visual analog scale (0-100 mm, with 0 indicating no pain and 100 indicating the worst pain).
Health Assessment Questionnaire-Disability Index (HAQ-DI) | A-319 within 1 year after subcutaneous injection (Day 15, Day 28, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12)
  The Health Assessment Questionnaire-Disability Index (HAQ-DI) is a component of the ACR evaluation and is also used to assess treatment efficacy. The HAQ-DI is a patient questionnaire assessing RA-related disability (physical function assessment). It consists of 20 questions across eight dimensions. Scaled on a 0-3 scale, 0 = no difficulty, 1 = some difficulty, 2 = very difficult, and 3 = unable to complete.
Simple Disease Activity Index (SDAI) | A-319 within 1 year after subcutaneous injection (Day 15, Day 28, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12)
  The Simple Disease Activity Index (SDAI) is a tool for assessing disease activity that integrates physical examination, acute reaction substances, patient reports, and physician assessments. It includes the following: swollen joints (0-28), tender joints (0-28), CRP (0.1-10 mg/dL), PaGA (0-100 mm), and PhGADA (0-100 mm).
Clinical Disease Activity Index (CDAI) | A-319 within 1 year after subcutaneous injection (Day 15, Day 28, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12)
  The Clinical Disease Activity Index (CDAI) is similar to the SDAI. This scale does not include laboratory tests and can be assessed immediately. The CDAI includes the following: swollen joints (0-28), tender joints (0-28), PaGA (0-100 mm), and PhGADA (0-100 mm).

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No